CLINICAL TRIAL: NCT02184715
Title: The Additional Therapeutic Effects of Virtual Reality System in Children With Developmental Delays
Brief Title: Effects of Virtual Reality System in Children With Developmental Delays
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ru-Lan Hsieh (Other)
Responsible Party: Sponsor-Investigator, Ru-Lan Hsieh, MD, Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: HP-01
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Developmental Delays
Keywords: virtual reality system, children, developmental delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual reality video game (Active Comparator): Participants received rehabilitation treatment and additional virtual reality system (30 minutes of interactive virtual reality system play, two times per week, in eight sessions over a 4-week span) for 1 month, followed by rehabilitation treatment for 1 month
  Interventions: Other: virtual reality system
- Virtual reality system (Placebo Comparator): received rehabilitation treatment for 1 month, followed by rehabilitation treatment and additional virtual reality system (30 minutes of interactive video game play, two times per week, in eight sessions over a 4-week span) during the one month of intervention period.
  Interventions: Other: virtual reality system

INTERVENTIONS:
Other: virtual reality system — The participants were randomly assigned to either Group A or Group B. Group A received rehabilitation treatment and additional virtual reality system for 1 month, followed by rehabilitation treatment for 1 month; by contrast, the participants in Group B received rehabilitation treatment for 1 month, followed by rehabilitation treatment and additional virtual reality system for 1 month.

SUMMARY:
The purpose of this study is to investigate the effects of virtual reality system on children with developmental delays.

DETAILED DESCRIPTION:
Participants attended eight 30-minute sessions of virtual reality system for 4 weeks in addition to regular rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* confirmed to have developmental delays
* provided informed consent
* 2 to 12 years old

Exclusion Criteria:

* failed to provide informed consent

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
health of children (Pediatric Quality of Life Inventory) | changes from baseline at one and two months.
  Following the recruitment and baseline assessment, outcome measures were assessed before treatment (Time 0), at the end of first intervention in the fourth week (Time 1), and at the end of second intervention in the eighth week (Time 2).

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital; Taipei Medical University
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsieh RL, Lee WC, Lin JH. The Impact of Short-Term Video Games on Performance among Children with Developmental Delays: A Randomized Controlled Trial. PLoS One. 2016 Mar 16;11(3):e0149714. doi: 10.1371/journal.pone.0149714. eCollection 2016. PMID 26983099